CLINICAL TRIAL: NCT06927167
Title: The Effect of Chin Tuck Exercises and Cervical Extension Exercises on Forward Head Posture
Brief Title: Effect of Exercises on Forward Head Posture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC-01008 Muhammad Haris
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Postural; Defect
Keywords: Forward Head Posture, chin tuck exercises.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chin tuck exercises (Experimental): Participants will perform supervised chin tuck exercises targeting deep cervical flexors
  Interventions: Other: Chin Tuck Exercise
- Seated cervical extension exercises (Experimental): Perform seated cervical extension exercises focusing on activating posterior neck muscles
  Interventions: Other: Seated cervical extension exercises

INTERVENTIONS:
Other: Chin Tuck Exercise — Chin Tuck Exercises and Cervical Extension Exercises on Forward Head Posture
  Arms: Chin tuck exercises
Other: Seated cervical extension exercises — Perform seated cervical extension exercises focusing on activating posterior neck muscles
  Arms: Seated cervical extension exercises

SUMMARY:
The Study aims to evaluate the effectiveness of chin tuck exercises in improving forward head posture.

To assess the impact of cervical extension exercises on forward head posture. To determine which exercise protocol provides superior results for FHP

DETAILED DESCRIPTION:
The study focus on understanding Forward head posture (FHP). Forward head posture (FHP) is a common musculoskeletal disorder characterized by a shift of the head forward in relation to the vertical axis of the body. This condition increases the load on the cervical spine, causing discomfort, pain and impaired musculoskeletal function. The incidence of FHP has increased significantly due to sedentary lifestyles and prolonged use of electronic devices, making it a pressing problem for healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Adults aged 30-45 years with diagnosed forward head posture.
* Chronic nonspecific neck pain for at least 3 months.
* FHP diagnosed via craniovertebral angle measurement.

Exclusion Criteria:

* Participants fall in this category would be excluded of the study.
* History of cervical spine surgery or trauma.
* Severe cervical instability or neurological deficits.
* Systemic diseases affecting posture.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral angle measurement | 4 weeks
  The craniovertebral angle (CVA) is a measurement of the angle between the neck and the head. It's used to assess head posture and forward head posture (FHP)

SECONDARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) for pain. | 4 weeks
  A Numerical Pain Rating Scale (NPRS) is a pain assessment tool where patients rate their pain intensity on a scale from 0 to 10, with "0" representing "no pain" and "10" representing "the worst pain imaginable

OTHER OUTCOMES:
Neck Disability Index (NDI) for functional outcomes. | 4 weeks
  The Neck Disability Index (NDI) is a questionnaire that measures how neck pain affects a person's daily life. It's used to assess functional outcomes and disability in patients with neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Ataur Rahman, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University malakand campus, Malakand, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No